CLINICAL TRIAL: NCT00093145
Title: A Phase II Study of Weekly Dose-Dense Nanoparticle Paclitaxel (ABI-007), Carboplatin With Herceptin® As First-Line Therapy of Advanced HER-2 Positive Breast Cancer
Brief Title: Study of Albumin-bound Paclitaxel (Abraxane) in Combination With Carboplatin and Herceptin in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA016; NCT00085605 (obsolete NCT alias)
Record Dates: First submitted 2004-10-04; First posted 2004-10-05 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Carboplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albumin-bound paclitaxel, Carboplatin + Herceptin (Experimental): Participants received albumin-bound paclitaxel, 100 mg/m^2 weekly every 3 out of 4 weeks, carboplatin at an area under the curve (AUC) = 6 every 4 weeks and Herceptin weekly, 4 mg/kg the first week and 2 mg/kg on all subsequent weeks by intravenous (IV) infusion for up to 6 cycles in the absence of disease progression or intolerable toxicity. Participants could continue treatment with chemotherapy beyond 6 cycles at the discretion of the investigator, but Herceptin therapy was to continue to be administered weekly (2 mg/kg) until intercurrent illness, disease progression, unacceptable toxicity, patient withdrawal or administration of any non-protocol anti-cancer treatment.
  Interventions: Drug: Albumin-bound paclitaxel; Drug: Carboplatin; Drug: Herceptin®

INTERVENTIONS:
Drug: Albumin-bound paclitaxel — Administered by intravenous infusion.
  Other Names: ABI-007; ABRAXANE®
Drug: Carboplatin — Carboplatin dose was calculated using a modified Calvert formula (creatinine clearance was substituted for GFR): Total dose (mg) = (target AUC) x (creatinine clearance + 25). Note: AUC = 6 was initially targeted, but could be decreased due to toxicity.
  Other Names: Paraplatin®
Drug: Herceptin® — Administered by IV infusion
  Other Names: Trastuzumab

SUMMARY:
This trial will treat patients with advanced breast cancer with a new anti-cancer medicine used in combination with two existing anti-cancer medications: Albumin-bound paclitaxel (ABI-007), Carboplatin and Herceptin. Participants will be given the combination therapy on a weekly basis and may continue on therapy as long as their condition improves and drug toxicity is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenocarcinoma of the breast
* Tumor shows 3+ overexpression of the human epidermal growth factor receptor 2 (HER-2)/proto-oncogene by immunohistochemistry assay, or is fluorescence in situ hybridization (FISH)+
* Stage IV disease
* Measurable disease
* At least 3 weeks since prior cytotoxic chemotherapy
* At least 4 weeks since radiotherapy with full recovery
* At least 4 weeks since major surgery with full recovery
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least 18 years old
* Absolute neutrophil count (ANC) at least 1.5 x 10^9 cells/L
* Platelets at least 100 x 10^9 cells/L
* Hemoglobin at least 9 g/dL
* Aspartame aminotransferase (AST), alanine aminotransferase (ALT) less than 2.5X upper limit normal
* Alkaline Phosphatase less than 1.5X upper limit normal
* Creatinine less than 1.5 gm/dL
* Normal left ventricular ejection fraction
* Negative pregnancy test
* Agree to use method to avoid pregnancy
* Informed Consent is obtained

Exclusion Criteria:

* Up to one regimen of prior neo-adjuvant or adjuvant chemotherapy is allowed. One year since Taxane and Herceptin treatment.
* Cumulative life-time dose of doxorubicin is greater than 360 mg/m^2
* Concurrent immunotherapy or hormonal therapy
* Parenchymal brain metastases, if present, must be documented to be clinically and radiographically stable for at least 6 months after treatment
* Serious intercurrent medical or psychiatric illness, including serious active infection
* History of congestive heart failure
* History of other malignancy within the last 5 years which could affect the diagnosis or assessment of breast cancer
* Patients who have received an investigational drug within the previous 3 weeks
* Patient is currently enrolled in another clinical study receiving investigational therapies
* Pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-06-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2008-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (14):
  - Breastlink Med Group, Long Beach, California
  - Hematology/Oncology P.C. Carl & Dorothy Bennet Cancer Center, Stamford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lombardi Cancer Center Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Cancer Institute, Hudson, Florida
  - Gulf Coast Oncology Associates, St. Petersburg, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Gerogia Cancer Specialist, Atlanta, Georgia
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Southwest Regional Cancer Center, Austin, Texas
  - Swedish Medical Center Cancer Institute Research, Seattle, Washington

REFERENCES:
- [Result] Conlin AK, Seidman AD, Bach A, Lake D, Dickler M, D'Andrea G, Traina T, Danso M, Brufsky AM, Saleh M, Clawson A, Hudis CA. Phase II trial of weekly nanoparticle albumin-bound paclitaxel with carboplatin and trastuzumab as first-line therapy for women with HER2-overexpressing metastatic breast cancer. Clin Breast Cancer. 2010 Aug 1;10(4):281-7. doi: 10.3816/CBC.2010.n.036. PMID 20705560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to slow patient accrual, only 32 patients of the planned 50 patients were enrolled. Patients were enrolled between June 2004 and July 2007.
Period: Overall Study
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Started | 32
At Least One Response Assessment | 31
Completed | 15 (Treatment completed upon progressive disease)
Not Completed | 17
Not completed — Unacceptable Toxicity Only | 2
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 9
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 52.0 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black, of African Heritage | 4
  White, Non-Hispanic and Non-Latino | 26
  White, Hispanic or Latino | 2
Region of Enrollment [Number; unit: participants]
  United States | 32
Menopausal Status [Number; unit: participants]
  Pre-Menopausal | 7
  Post-Menopausal | 25
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale used to assess the progress of disease, how the disease affects the daily living abilities of the patient, and to determine appropriate treatment and prognosis.
  0=Fully active, able to perform all pre-disease activity. 1=Restricted in physically strenuous activity, ambulatory, able to perform light work. 2=Ambulatory, capable of all selfcare, unable to carry out any work activities. Up and about >50% of waking hours. 3=Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4=Completely disabled. Cannot perform any selfcare. Confined to bed or chair. 5=Dead.
  participants
    0 (Fully Active) | 19
    1 (Restrictive but Ambulatory) | 12
    2 (Ambulatory, but Unable to Work) | 1
Physician assessment of peripheral neuropathy [Number; unit: participants] — The physician assessed sensory neuropathy using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) of "Neurology -- Neuropathy - Sensory". The scale is 0=normal and 1=asymptomatic; loss of deep tendon reflexes or paresthesia (including tingling) but not interfering with function. Data available for 31 participants.
  participants
    Grade 0 | 30
    Grade 1 | 1
Histology of Primary Diagnosis [Number; unit: participants]
  Carcinoma/Adenocarcinoma | 31
  Other | 1
Time from first documented metastatic disease to study entry [Median (Full Range); unit: years] | 0.1 [0 to 6]
Specific site(s) of metastasis/relapse [Number; unit: participants] — Participants can be in multiple sites of metastasis/relapse categories.
  participants
    Brain/Central Nervous System | 1
    Skin/Soft Tissue/Breast | 21
    Lymph Nodes | 24
    Lung | 19
    Liver | 15
    Peritoneal | 1
    Bone | 22
    Other | 1
Dominant site of metastasis/relapse [Number; unit: participants]
  Visceral | 24
  Non Visceral | 8
Number of Lesions (Target + Non-Target) [Number; unit: participants]
  0 or 1 lesion | 0
  2 to 3 lesions | 10
  > 3 lesions | 22
Dominant Lesion Site (Target + Non-Target) [Number; unit: participants]
  Visceral | 25
  Non visceral | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Objective Confirmed Complete or Partial Overall Response
Description: Percentage of participants who achieved an objective confirmed complete or partial overall response based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. A complete response (CR) is the disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation. A partial response (PR) is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 4 weeks after initial documentation. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing, or with the persistence of one or more non-target lesions and/or the maintenance of tumor marker level above the normal limits.
Time Frame: Objective response was evaluated every 2 cycles, up to a maximum of 39 cycles (approximately 39 months)
Population: The treated population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 32
Percentage of participants | 62.5 [45.7 to 79.3]

2. Secondary Outcome: Percentage of Participants With a Total Response
Description: Total response was defined as the percentage of participants with stable disease (SD) for ≥ 16 weeks or complete or partial overall response. Stable disease was defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease. Progressive disease is at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: Evaluated every 2 cycles, up to a maximum of 39 cycles.
Population: Treated population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 32
percentage of participants | 81.3 [67.7 to 94.8]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was measured from the date of first dose of study drug to the start of disease progression. Patients who did not have disease progression at the end of follow-up were censored at the last known time that the patient was evaluated for progression. Progression is at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion. Time to disease progression was summarized using Kaplan-Meier methods.
Time Frame: Assessed every 2 cycles, up to a maximum of 39 cycles.
Population: Treated population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 32
months | 16.6 [7.5 to 26.5]

4. Secondary Outcome: Duration of Response
Description: Duration of response was evaluated by measuring progression-free survival for participants with a complete response or partial response. Progression-free survival was defined as the time from the first dose of study drug to the start of progression or patient death (whichever occurred first). Participants who did not have progression or were still alive were censored at the last known time the patient was progression free. Patients that initiated other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated. Progression is at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: Assessed every 2 cycles, up to a maximum of 39 cycles.
Population: Treated Population - Patients with a Confirmed Complete or Partial Overall Response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 20
months | 17.8 [15.9 to 37.0]

5. Secondary Outcome: Overall Patient Survival
Description: Overall survival was defined as the time from the day of randomization to patient death (due to any cause), as assessed by post study follow-up on a monthly basis for 3 months and every 3 months. Participants still alive were censored at the last known time that the patient was alive. Patient survival was estimated using Kaplan-Meier methods.
Time Frame: From Day 1 until approximately 44 months.
Population: Treated population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 32
months | NA [NA to NA] — Overall survival could not be estimated due to the low number of deaths.

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A Treatment-emergent AE was any AE that began or worsened after the start of study drug through 30 days after the last dose of study drug or end of study whichever is later. A treatment related toxicity was one considered by the investigator to be possibly, probably or definitely related to study drug. AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE) on the following scale: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death. A serious adverse event (SAE) is any untoward medical occurrence at any dose that: is fatal or life-threatening; results in persistent or significant disability or incapacity; requires or prolongs in-patient hospitalization; is a congenital anomaly/birth defect in the offspring of a patient; and conditions not included in the above that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above
Time Frame: Day 1 up to 39 cycles
Population: Treated population
Measure: Number; unit: participants
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Number analyzed (Participants) | 32
participants
  Number with any treatment emergent AE | 32
  Number with any treatment-related AE | 31
  Number with any Grade 3/4 TEAE | 20
  Number with any serious AE | 5

ADVERSE EVENTS:
Time Frame: Day 1 up to 39 months
Arm/Group | Albumin-bound Paclitaxel, Carboplatin + Herceptin
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-bound Paclitaxel, Carboplatin + Herceptin (N=32)
Hypersensitivity (Immune system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Catheter site infection (Infections and infestations) | 1
Confusional state (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-bound Paclitaxel, Carboplatin + Herceptin (N=32)
Nausea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 27
Pyrexia (General disorders) | 8
Pain (General disorders) | 7
Rigors (General disorders) | 7
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 4
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Performance status decreased (General disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 21
Anaemia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 14
Headache (Nervous system disorders) | 9
Neuropathy (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Facial pain (Musculoskeletal and connective tissue disorders) | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Insomnia (Psychiatric disorders) | 17
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 6
Alanine aminotransferase increased (Investigations) | 6
White blood cell count decreased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 3
Weight decreased (Investigations) | 3
White blood cell count (Investigations) | 3
Blood creatinine abnormal (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 9
Acne (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypersensitivity (Immune system disorders) | 3
Drug hypersensitivity (Immune system disorders) | 4
Hypertension (Vascular disorders) | 4
Lymphoedema (Vascular disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Vision blurred (Eye disorders) | 4
Breast pain (Reproductive system and breast disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Tachycardia (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Sponsor a copy of the manuscript at least 30 days prior to submission; if no response is received within 30 days the publication or presentation may proceed without delay. Sponsor may request that Confidential Information be deleted. Publication may be delayed for an additional 60 days if patentable matter is included.